CLINICAL TRIAL: NCT05144815
Title: Effectiveness of an Endurance Exercise Programme Preceded by Ischaemic Preconditioning in Older People: a Randomised Clinical Trial
Brief Title: Effectiveness of an Endurance Exercise Programme Preceded by Ischaemic Preconditioning in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151121
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Older People

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC + Exercise protocol group (Experimental): Patients in this group (n=16) will undergo ischaemic preconditioning (IPC) plus an endurance training protocol.
  Interventions: Other: IPC + Exercise protocol
- Sham IPC + Exercise protocol group (Sham Comparator): Patients in this group (n=16) will undergo sham ischaemic preconditioning (IPC) plus an endurance training protocol.
  Interventions: Other: Sham IPC + Exercise protocol

INTERVENTIONS:
Other: IPC + Exercise protocol — The intervention consists of two parts: IPC and endurance training protocol.
  IPC: participants will be placed in a supine position and a pneumatic compression cuff (Riester Komprimeter, Jungingen Germany) (96 centimetres long x 13 centimetres wide) will be placed on the proximal part of each lower extremity. Occlusion will then be performed by inflating the cuff to 220 mmHg for 5 minutes, followed by reperfusion to 0 mmHg for 5 minutes. Each session will consist of 3 sets of 5 minutes of ischaemia followed by 5 minutes of reperfusion.
  Endurance training protocol: walking 20 min at moderate intensity (i.e. 64- 76 % HRmax, 12-13 Borg Scale) in a circuit designed in an open field, 3 times a week, for 6 weeks.
  Arms: IPC + Exercise protocol group
Other: Sham IPC + Exercise protocol — The intervention consists of two parts: sham IPC and endurance training protocol.
  Sham IPC: the pressure cuff will be inflated by only 10 mmHg, so that it will act as a placebo.
  Endurance training protocol: walking 20 min at moderate intensity (i.e. 64- 76 % HRmax, 12-13 Borg Scale) in a circuit designed in an open field, 3 times a week, for 6 weeks.
  Arms: Sham IPC + Exercise protocol group

SUMMARY:
In recent decades, the proportion of people over 65 years of age is increasing rapidly, due to rising life expectancy and declining fertility rates. According to the World Health Organization, people in this age group will constitute 22% of the population by 2050, up from the current 12% (WHO, 2018). Therefore, improving quality of life (healthspan) and preventing disability has become a public health challenge (Olshansky, 2018).

In this context, physical exercise has been shown to be able to prevent sarcopenia, functional decline, the presence of chronic diseases and even mortality in this group (Izquierdo et al., 2021; Lazarus, Lord, & Harridge, 2019).

A training method that could enhance the benefits of walking is ischaemic preconditioning (IPC), characterised by the application of brief periods of circulatory occlusion-reperfusion to a limb, minutes to hours prior to exercise. This type of intervention, initially used to delay/prevent cell damage in patients with myocardial infarction (Murry, Jennings, & Reimer, 1986), has recently shown beneficial effects in young people to improve physical performance in a wide variety of sports (Caru, Levesque, Lalonde, & Curnier, 2019), as well as to improve recovery from associated muscle damage (Franz et al., 2018), which is of particular interest in the adult population. In fact, the application of IPC alone for two weeks has been shown to improve walking speed and reduce fatigue in post-stroke patients (Durand et al., 2019), promising effects that could be increased when applied prior to resistance training, such as walking.

Thus, the objective of this study is to determine the effectiveness of an endurance exercise programme preceded by ischaemic preconditioning on parameters related to physical function, cognitive status and quality of life in older people. In addition, we set out to compare the acute and chronic effect of the proposed interventions.

DETAILED DESCRIPTION:
In recent decades, the proportion of people over 65 years of age is increasing rapidly, due to rising life expectancy and declining fertility rates. According to the World Health Organization, people in this age group will constitute 22% of the population by 2050, up from the current 12% (WHO, 2018). Therefore, improving quality of life (healthspan) and preventing disability has become a public health challenge (Olshansky, 2018).

In this context, physical exercise has been shown to be able to prevent sarcopenia, functional decline, the presence of chronic diseases and even mortality in this group (Izquierdo et al., 2021; Lazarus, Lord, & Harridge, 2019).

Resistance or endurance training can improve sarcopenia, reduce intramuscular fat accumulation, improve muscle function, among others. Aerobic exercise has been shown to be effective in maintaining muscle mass and strength in older adults is walking (Kubo et al., 2008). In fact, walking can also improve VO2max in older adults when intensities are above ∼40% VO2max (Nemoto, Gen-no, Masuki, Okazaki, & Nose, 2007). In addition, it has been linked to the prevention of cognitive decline (Maki et al., 2012) and improvements in quality of life (Awick et al., 2015) in older people.

A training method that could enhance the benefits of walking is ischaemic preconditioning (IPC), characterised by the application of brief periods of circulatory occlusion-reperfusion to a limb, minutes to hours prior to exercise. This type of intervention, initially used to delay/prevent cell damage in patients with myocardial infarction (Murry, Jennings, & Reimer, 1986), has recently shown beneficial effects in young people to improve physical performance in a wide variety of sports (Caru, Levesque, Lalonde, & Curnier, 2019), as well as to improve recovery from associated muscle damage (Franz et al., 2018), which is of particular interest in the adult population. In fact, the application of IPC alone for two weeks has been shown to improve walking speed and reduce fatigue in post-stroke patients (Durand et al., 2019), promising effects that could be increased when applied prior to resistance training, such as walking.

Thus, the objective of this study is to determine the effectiveness of an endurance exercise programme preceded by ischaemic preconditioning on parameters related to physical function, cognitive status and quality of life in older people. In addition, we set out to compare the acute and chronic effect of the proposed interventions.

Therefore, this study is a randomized clinical trial in which three groups of twenty people in each group will participate, with different interventions:

* Experimental group 1: Exercise protocol + IPC.
* Experimental group 2: Exercise protocol + sham IPC.
* Control group. Participants will be evaluated in four moments, at baseline, immediately after the first session, postintervention (after 6-week intervention) and 4-week follow-up.

Data analysis will be performed with SPSS statistic program (v26). Normality and homoscedasticity will be analyzed by Shapiro-Wilk t-test and Levene test, respectively. For comparation between groups Bonferroni will be used. If any confusion factor that not meet requirements to be analysed like a covariable exist, ANCOVA will be used. When p<0.0.5 statistical significant differences will be assumed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 -90 years
* Physically inactive (< 150 minutes of physical activity per week).
* Signed informed consent form

Exclusion Criteria:

* Institutionalised patients.
* History of stroke in the last 6 months or hospital admission for any reason in the last 3 months.
* Uncontrolled hypertension.
* Medication with anticoagulants.
* Oncological patient with active treatment: chemotherapy or radiotherapy.
* Neurological or cardiovascular musculoskeletal pathology that contraindicates physical activity.
* Cognitive impairment (score below 25 on the "Mini-mental Test"); or severe disability (score below 15 points on the Barthel scale).
* Completion of less than 80% of training sessions.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 8 minutes
  "6 minutes walking test" (6MWT)
Heart rate variability during walking | 40 minutes
  Heart rate monitor RS800CX (Polar Electro Oy Kempele, Finland).

SECONDARY OUTCOMES:
Lower limb strength: for the assessment of isometric strength | 10 minutes
  A load cell (CTCS; Mutronic) will be used to measure the strength of the intrinsic and extrinsic muscles of the hip, knee and ankle
Muscle mass (sacopenia) | 3 minutes
  Bioimpedance (Tanita DC-430MA, Tanita Corporation of America, Inc., Arlington Heights, IL, USA).
General physical condition | 5 minutes
  Short Physical Performance Battery
Fatigue | 1 minute
  Borg scale 20
Fall risk, agility and dynamic balance | 3 minutes
  Fall skip
Independence in basic activities of daily living (BADL) and instrumental activities of daily living (IADL) | 5 minutes
  Barthel Index and Lawton and Brody scale, respectively
Health-related Quality of Life | 2 minutes
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Marta Inglés, Dr, Principal Investigator — Univeristy of Valencia
Locations (2):
- Spain (2):
  - Elena Muñoz, Valencia, Valencia / València
  - Marta Inglés, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Nemoto K, Gen-no H, Masuki S, Okazaki K, Nose H. Effects of high-intensity interval walking training on physical fitness and blood pressure in middle-aged and older people. Mayo Clin Proc. 2007 Jul;82(7):803-11. doi: 10.4065/82.7.803. PMID 17605959
- [Background] Ziaaldini MM, Koltai E, Csende Z, Goto S, Boldogh I, Taylor AW, Radak Z. Exercise training increases anabolic and attenuates catabolic and apoptotic processes in aged skeletal muscle of male rats. Exp Gerontol. 2015 Jul;67:9-14. doi: 10.1016/j.exger.2015.04.008. Epub 2015 Apr 21. PMID 25910622
- [Derived] Munoz-Gomez E, Molla-Casanova S, Sempere-Rubio N, Serra-Ano P, Aguilar-Rodriguez M, Moreno-Segura N, Chulvi-Medrano I, Ingles M. Effectiveness of an endurance exercise programme preceded by ischaemic preconditioning in older people. Geriatr Nurs. 2025 May-Jun;63:442-449. doi: 10.1016/j.gerinurse.2025.03.043. Epub 2025 Apr 18. PMID 40252516